CLINICAL TRIAL: NCT05198492
Title: Short- and Long-term Health Effects of Air Pollution in Poland
Acronym: EP-PARTICLES
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Collaborators: Charles University, Czech Republic (Other); University of Liverpool (Other); University of Skopje (Other); University of Lodz (Unknown)
Responsible Party: Principal Investigator, Lukasz Kuzma, Principal Investigator, Medical University of Bialystok
Other Study IDs: UMB-KKI-104
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Acute Coronary Syndrome; Atrial Fibrillation; Kidney Diseases; Particulate Matter Inhalation Injury; Pollution; Exposure; Oxidative Stress; Ischemic Stroke
Keywords: Air Pollution; Public Health; Acute Coronary Syndromes; Atrial Fibrillation; Kidney Diseases; Particulate Matter; Cardiovascular Diseases
MeSH Terms: conditions — Acute Coronary Syndrome; Atrial Fibrillation; Kidney Diseases; Ischemic Stroke; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Patients with hospitalizations or emergency room visits due to acute coronary syndromes: Data on hospitalization for acute coronary syndromes were obtained and extracted from the National Health Fund reports. In the present analysis, we used data from patients registered as residents in the Podlaskie, Lubelskie, Podkarpackie, Świetokrzyskie, and Warminsko-Mazurskie voivodeships from January 1, 2011 to December 31, 2020. The set of variables that were subjected to the analysis included demographic features and ICD-10 codes. The diagnosis was based on reports obtained from to the National Health Fund, and these reports have not been reviewed with patient hospital documentation.
  Interventions: Other: Impact of air pollution
- Patients with hospitalizations or emergency room visits due to atrial fibrillation: Data on hospitalization for atrial fibrillation were obtained and extracted from the National Health Fund reports. In the present analysis, we used data from patients registered as residents in the Podlaskie, Lubelskie, Podkarpackie, Świetokrzyskie, and Warminsko-Mazurskie voivodeships from January 1, 2011 to December 31, 2020. The set of variables that were subjected to the analysis included demographic features and ICD-10 codes. The diagnosis was based on reports obtained from to the National Health Fund, and these reports have not been reviewed with patient hospital documentation.
  Interventions: Other: Impact of air pollution
- Patients with hospitalizations or emergency room visits due to kidney diseases: Data on hospitalization for kidney diseases were obtained and extracted from the National Health Fund reports. In the present analysis, we used data from patients registered as residents in the Podlaskie, Lubelskie, Podkarpackie, Świetokrzyskie, and Warminsko-Mazurskie voivodeships from January 1, 2011 to December 31, 2020. The set of variables that were subjected to the analysis included demographic features and ICD-10 codes. The diagnosis was based on reports obtained from to the National Health Fund, and these reports have not been reviewed with patient hospital documentation.
  Interventions: Other: Impact of air pollution
- Patients who died due to cardiovascular diseases: Data on mortality were collected from the National Statistical Office in Poland. These include information on all the deaths recorded in the Podlaskie, Lubelskie, Podkarpackie, Świetokrzyskie, and Warminsko-Mazurskie voivodeships from January 1, 2011 to December 31, 2020 The records included sex and age of people who had died, and the causes of deaths were classified according to codes in the International Classification of Diseases-10th Revision (ICD-10).
  Interventions: Other: Impact of air pollution
- Patients who died due to neoplasm diseases: Data on mortality were collected from the National Statistical Office in Poland. These include information on all the deaths recorded in the Podlaskie, Lubelskie, Podkarpackie, Świetokrzyskie, and Warminsko-Mazurskie voivodeships from January 1, 2011 to December 31, 2020 The records included sex and age of people who had died, and the causes of deaths were classified according to codes in the International Classification of Diseases-10th Revision (ICD-10).
  Interventions: Other: Impact of air pollution
- Patients who died due to kidney diseases: Data on mortality were collected from the National Statistical Office in Poland. These include information on all the deaths recorded in the Podlaskie, Lubelskie, Podkarpackie, Świetokrzyskie, and Warminsko-Mazurskie voivodeships from January 1, 2011 to December 31, 2020 The records included sex and age of people who had died, and the causes of deaths were classified according to codes in the International Classification of Diseases-10th Revision (ICD-10).
  Interventions: Other: Impact of air pollution
- Patients with hospitalizations or emergency room visits due to ischemic strokes: Data on hospitalization for ischemic strokes were obtained and extracted from the National Health Fund reports. In the present analysis, we used data from patients registered as residents in the Podlaskie, Lubelskie, Podkarpackie, Świetokrzyskie, and Warminsko-Mazurskie voivodeships from January 1, 2011 to December 31, 2020. The set of variables that were subjected to the analysis included demographic features and ICD-10 codes. The diagnosis was based on reports obtained from to the National Health Fund, and these reports have not been reviewed with patient hospital documentation.
  Interventions: Other: Impact of air pollution

INTERVENTIONS:
Other: Impact of air pollution — To assess the short- and long- term impact of air pollution

SUMMARY:
The effects of air pollution on the frequency of hospital admissions and mortality due to acute coronary syndromes, atrial fibrillation, and renal disfunction are noted also in areas perceived as pollution-free (due to the lack of large industry). The aim of the project is to assess the impact of air pollution in Eastern Poland on regional public health.

DETAILED DESCRIPTION:
The project will be conducted in Eastern Poland - the area characterized by unique natural features, large areas covered by forests, lack of factories, and relatively low industrialization. On the other hand, the region is also characterized by low socioeconomic status, in the cold season the residents' suboptimal heating choices are in result posing a major anthropogenic threat to air quality in the form of low emissions. The vast majority of studies on air pollution were conducted in highly polluted areas, in which patients are exposed to moderate and extreme concentrations of pollutants. Taking into consideration the scarce number of surveys from areas with a low level of pollution the investigators intend to analyze the relationship between air pollution and cardiovascular and renal outcomes in Eastern Poland. The examination of the impact of so-called "Polish smog" on mortality and morbidity in the study area is not without significance. It would be the first major study of the impact of this type of pollution on human health.

In the subsequent part of the study, we will evaluate the effects of Polish smog in the entire country.

In light of extant body of literature, the following will be considered as the public health indicators: acute coronary syndromes, episodes of atrial fibrillation, ischemic strokes, kidney disease hospitalizations or emergency room visits, cardiovascular and renal mortality.

ELIGIBILITY:
Inclusion Criteria:

* Residents from the analyzed area

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be based on residents of Eastern Poland. This term covers 5 voivodships - Warmińsko-Mazurskie, Podlaskie, Lubelskie, Świętokrzyskie, Podkarpackie - with total area of 99,004 km2. The inhabitants of this region constitute 21.3% of the population of Poland and 1.6% of the population of the European Union. The area characterized by unique natural features, large areas covered by forests, lack of factories, and relatively low industrialization is not free of air pollution. As the region is also characterized by low socioeconomic status, in the cold season the residents' suboptimal heating choices are in result posing a major anthropogenic threat to air quality in the form of low emissions.
Sampling Method: Non-Probability Sample
Enrollment: 8300000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of acute coronary syndromes related to the impact of air pollution. | Through study completion, an average of 1 year
  Short- and long- term influence of air pollution on the number of hospital admissions for acute coronary syndromes.
Number of atrial fibrillation episodes related to the impact of air pollution. | Through study completion, an average of 1 year
  Short- and long- term influence of air pollution on the number of hospital admissions for atrial fibrillation.
Number of hospitalizations due to kidney diseases related to the impact of air pollution. | Through study completion, an average of 1 year
  Long- term influence of air pollution on the number of hospital admissions for kidney disease.
Number of hospitalizations due to acute kidney diseases related to the impact of air pollution. | Through study completion, an average of 1 year
  Long- term influence of air pollution on the number of hospital admissions for kidney disease.
Number of patients under hemodialysis related to the impact of air pollution. | Through study completion, an average of 1 year
  Long- term influence of air pollution on the number of hospital admissions for kidney disease.
Number of ischemic strokes related to the impact of air pollution. | Through study completion, an average of 1 year
  Short- and long- term influence of air pollution on the number of hospital admissions for ischemic strokes.

SECONDARY OUTCOMES:
Cardiovascular mortality | Through study completion, an average of 1 year
  Short- and long- term influence of air pollution on the number of cardiovascular mortality.
Neoplasm mortality | Through study completion, an average of 1 year
  Short- and long- term influence of air pollution on neoplasm mortality.
Kidney disease mortality | Through study completion, an average of 1 year
  Short- and long- term influence of air pollution on mortality related to renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Kuźma, Study Director — Medical University of Bialystok
Locations (1):
- Department of Invasive Cardiology, Medical University of Bialystok, Bialystok, Podlaskie Voivodeship, Poland

REFERENCES:
- [Background] Kuzma L, Dabrowski EJ, Kurasz A, Bachorzewska-Gajewska H, Dobrzycki S. The 10-Year Study of the Impact of Particulate Matters on Mortality in Two Transit Cities in North-Eastern Poland (PL-PARTICLES). J Clin Med. 2020 Oct 27;9(11):3445. doi: 10.3390/jcm9113445. PMID 33120927
- [Background] Kuzma L, Struniawski K, Pogorzelski S, Bachorzewska-Gajewska H, Dobrzycki S. Gender Differences in Association between Air Pollution and Daily Mortality in the Capital of the Green Lungs of Poland-Population-Based Study with 2,953,000 Person-Years of Follow-Up. J Clin Med. 2020 Jul 23;9(8):2351. doi: 10.3390/jcm9082351. PMID 32717977
- [Background] Kuzma L, Malyszko J, Bachorzewska-Gajewska H, Kralisz P, Dobrzycki S. Exposure to air pollution and renal function. Sci Rep. 2021 Jun 1;11(1):11419. doi: 10.1038/s41598-021-91000-0. PMID 34075149
- [Background] Kuzma L, Wanha W, Kralisz P, Kazmierski M, Bachorzewska-Gajewska H, Wojakowski W, Dobrzycki S. Impact of short-term air pollution exposure on acute coronary syndrome in two cohorts of industrial and non-industrial areas: A time series regression with 6,000,000 person-years of follow-up (ACS - Air Pollution Study). Environ Res. 2021 Jun;197:111154. doi: 10.1016/j.envres.2021.111154. Epub 2021 Apr 17. PMID 33872649
- [Background] Kuzma L, Pogorzelski S, Struniawski K, Bachorzewska-Gajewska H, Dobrzycki S. Exposure to air pollution-a trigger for myocardial infarction? A nine-year study in Bialystok-the capital of the Green Lungs of Poland (BIA-ACS registry). Int J Hyg Environ Health. 2020 Aug;229:113578. doi: 10.1016/j.ijheh.2020.113578. Epub 2020 Aug 3. PMID 32758862
- [Background] Kuzma L, Pogorzelski S, Struniawski K, Dobrzycki S, Bachorzewska-Gajewska H. Effect of air pollution on the number of hospital admissions for acute coronary syndrome in elderly patients. Pol Arch Intern Med. 2020 Jan 31;130(1):38-46. doi: 10.20452/pamw.15064. Epub 2019 Nov 19. PMID 31742576
- [Result] Kuzma L, Dabrowski EJ, Kurasz A, Swieczkowski M, Jemielita P, Kowalewski M, Wanha W, Kralisz P, Tomaszuk-Kazberuk A, Bachorzewska-Gajewska H, Dobrzycki S, Lip GYH. Effect of air pollution exposure on risk of acute coronary syndromes in Poland: a nationwide population-based study (EP-PARTICLES study). Lancet Reg Health Eur. 2024 Apr 22;41:100910. doi: 10.1016/j.lanepe.2024.100910. eCollection 2024 Jun. PMID 38665621
- [Result] Swieczkowski M, Dobrzycki S, Kuzma L. Multi-City Analysis of the Acute Effect of Polish Smog on Cause-Specific Mortality (EP-PARTICLES Study). Int J Environ Res Public Health. 2023 Apr 18;20(8):5566. doi: 10.3390/ijerph20085566. PMID 37107848
- [Derived] Swieczkowski M, Lip GYH, Kurasz A, Jemielita P, Duzinkiewicz M, Januszko T, Dobrzycki S, Kuzma L. Short-term exposure to air pollution and risk of ischemic stroke requiring intravenous thrombolysis: a population-level analysis in Poland from the EP-PARTICLES study. Environ Health. 2025 Sep 29;24(1):69. doi: 10.1186/s12940-025-01230-2. PMID 41024000
- [Derived] Swieczkowski M, Lip GYH, Abohashem S, Jemielita P, Kurasz A, Duzinkiewicz M, Januszko T, Tomaszuk-Kazberuk A, Dobrzycki S, Kuzma L. Interplay between mental health, greenness, and environmental factors in cardiovascular mortality: insights from AIR-MIND. Eur J Prev Cardiol. 2025 Dec 23;32(18):1915-1927. doi: 10.1093/eurjpc/zwaf534. PMID 40884214
- [Derived] Swieczkowski M, Lip GYH, Kurasz A, Dabrowski EJ, Tomaszuk-Kazberuk A, Kaminski JW, Struzewska J, Dobrzycki S, Kuzma L. Association between exposure to air pollution and increased ischaemic stroke incidence: a retrospective population-based cohort study (EP-PARTICLES study). Eur J Prev Cardiol. 2025 Mar 18;32(4):276-287. doi: 10.1093/eurjpc/zwae301. PMID 39301834